CLINICAL TRIAL: NCT04095299
Title: Randomized Trial of Standard Dose Versus High Dose of Radiotherapy in Rectal Preservation With Chemo-radiotherapy to Patients With Early Low and Mid Rectal Cancer: The Watchful Waiting 3 Trial (WW3)
Brief Title: Standard Dose Versus High Dose of Radiotherapy in Rectal Preservation With Chemo-radiotherapy in Rectal Cancer Patients
Acronym: WW3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WW3
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Rectum
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Enrollment will continue until 162 patients have reached the primary endpoint two years after start of treatment. During these two years the total number of patients will therefore expectedly increase to approximately 290. This will be the population for secondary analyses and long-term follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Standard chemoradiotherapy (Active Comparator): 50.4 Gy to the tumor and elective volume. The dose is given in 28 fractions on weekdays concomitantly with capecitabine 825 mg/m2 twice daily on weekdays.
  Interventions: Radiation: 50.4 Gy to the tumor and elective volume; Drug: Capecitabine 825 mg/m2 twice daily on weekdays
- B: High-dose radiotherapy (Experimental): 62 Gy to the clinical tumor volume and 50.4 Gy to the elective volume. The dose is given in 28 fractions on weekdays concomitantly with capecitabine 825 mg/m2 twice daily on weekdays
  Interventions: Radiation: 62 Gy to the clinical tumor volume and 50.4 Gy to the elective volume; Drug: Capecitabine 825 mg/m2 twice daily on weekdays

INTERVENTIONS:
Radiation: 50.4 Gy to the tumor and elective volume — Standard radiotherapy
  Arms: A: Standard chemoradiotherapy
Radiation: 62 Gy to the clinical tumor volume and 50.4 Gy to the elective volume — Experimental radiotherapy
  Arms: B: High-dose radiotherapy
Drug: Capecitabine 825 mg/m2 twice daily on weekdays — Standard chemotherapy

SUMMARY:
In recent years, an increasing number of retrospective and prospective observational studies have indicated that a subset of rectal cancer patients may avoid surgery if they can achieve a complete response to chemoradiotherapy. Prospective trials, including the previous Danish Watchful Waiting trials (NCT00952926, NCT02438839) in early rectal cancer have demonstrated high levels of organ preservation with dose-escalation, but it is unclear whether this was primarily due to tumor stage or dose level.

The aim of the present study is to investigate if a higher dose of radiotherapy is superior compared to a standard dose in patients with early rectal cancer undergoing chemoradiotherapy with curative intent.

DETAILED DESCRIPTION:
The main curative treatment modality for rectal cancer is surgery, potentially combined with chemotherapy and radiotherapy to lower the risk of local recurrence. In recent years, an increasing number of retrospective and prospective observational studies have indicated that a subset of patients may avoid surgery altogether if they can achieve a complete response to chemoradiotherapy. These studies have mainly focused on locally advanced tumors with a high risk of local recurrence. Smaller, less advanced tumors appear to respond better to chemoradiotherapy, but the optimal treatment for non-surgical management has not been established. Prospective trials, including the previous Danish Watchful Waiting trials (NCT00952926, NCT02438839) in early rectal cancer have demonstrated high levels of organ preservation with dose-escalation, but it is unclear whether this was primarily due to tumor stage or dose level. High-level evidence is currently absent for the question of radiotherapy dose, especially in early stage cancers.

The aim of the present study is to investigate if a higher dose of radiotherapy is superior compared to a standard dose in patients with early rectal cancer undergoing chemoradiotherapy with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically verified adenocarcinoma of the rectum
* MDT conference finds patient a candidate for rectal resection
* Clinical tumor category cT1-3
* MRI findings

  * Maximal cross-sectional size of 4.5 cm (axial plane relative to the rectum)
  * Lowest edge of tumor located at or below the peritoneal reflection on MRI
* Performance status 0-2
* Age ≥ 18 years
* Eligible for radiotherapy and capecitabine according to investigator, including

  * Adequate function of bone marrow (neutrophils ≥ 1.5 x 10^9/l and thrombocytes ≥ 100 x 10^9/l)
  * Adequate function of liver (ALAT < 2.5 x upper limit of normal, bilirubin < 2.5 x upper limit of normal)
  * Adequate kidney function (Serum creatinine < 1.5 x upper limit of normal or measured GFR > 30 ml/min)
* Fertile women must present a negative pregnancy test and use secure contraceptives during and three months after treatment
* Written and orally informed consent

Exclusion Criteria:

* Previous surgical treatment of the present cancer, including transanal excision of tumor
* Other malignant disease within the past five years except non-melanoma skin cancer and premalignant lesions such as carcinoma in situ
* Distant metastases verified by imaging or biopsy, i.e. cM1
* Previous radiation treatment of the pelvis
* Pregnant or breastfeeding women.
* Existing colostomy or ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Rectal preservation at two years | 2 years after start of treatment
  * Presence of a full-length rectum, i.e. no rectal resection.
  * Absence of rectal tumor, malignant lymph nodes or any other tumor deposit or recurrence within the pelvis based on clinical examination, CT and MR
  * No stoma because of side effects to treatment or rectal dysfunction

SECONDARY OUTCOMES:
Rate of complete response within four months from start of radiotherapy | 4 months
Locoregional recurrence (within the pelvis) | At least yearly up to 5 years
Relapse free survival | At least yearly up to 5 years
Overall survival | At least yearly up to 5 years
Colostomy-free survival | At least yearly up to 5 years
Quality of life as assessed ny the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CR29+C30 | Up to 5 years
  QLQ is a 30-question assessment of quality of life. Twenty-eight questions are assessed on a scale of 1 (Not at all) to 4 (Very much); 2 questions are assessed on a scale of 1 (very poor) to 7 (excellent). Score range 0- 100. In the function scales, score 100 is best (more function). In the symptom scales, score 100 is worst, (more symptoms). The colorectal cancer module QLQ-CR29 should always be complemented by QLQ-C30. It contains four functional scales and 18 symptom scales. Some scales are dependent on gender and some are for patients with or without a stoma. There are 19 individual items assessed on a scale of 1 (Not at all) to 4 (Very much). Scores are totaled from each item to form the scales, and then normalized to 0-100.
Frequency of grade 3-4 toxicity according to CTCAE v4 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Jensen, MD, PhD, Principal Investigator — Department of Oncology, Vejle Hospital - University Hospital of Southern Denmark
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Copenhagen University Hospital, Righshospitalet and Bispebjerg Hospital, Copenhagen
  - Zealand University Hospital, Næstved, Næstved
  - Zealand University Hospital, Roskilde, Roskilde
  - Department of Oncology, Vejle Hospital, Vejle